CLINICAL TRIAL: NCT03370341
Title: Stimulating the Brain to Improve Self-Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Amy Pinkham, PhD, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-127
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will complete active and sham simulation sessions in a randomized, counterbalanced order approximately one week apart.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active anodal tDCS first, then Sham tDCS (Experimental): Active anodal tDCS (20 minutes) followed by behavioral testing; Washout (1 week); sham stimulation (20 minutes) followed by behavioral testing Intervention: Device: active anodal tDCS and sham tDCS
  Interventions: Device: active anodal tDCS; Device: sham tDCS
- Sham tDCS first, then Active anodal tDCS (Sham Comparator): Sham tDCS (20 minutes) followed by behavioral testing; Washout (1 week); Active anodal tDCS (20 minutes) followed by behavioral testing Intervention: Device: sham tDCS and sham tDCS
  Interventions: Device: active anodal tDCS; Device: sham tDCS

INTERVENTIONS:
Device: active anodal tDCS — active anodal tDCS with behavioral tasks to assess IA
Device: sham tDCS — sham tDCS with behavioral tasks to assess IA

SUMMARY:
This study investigates whether Introspective Accuracy (IA) can be improved in individuals with schizophrenia by stimulating the brain via transcranial Direct Current Stimulation (tDCS).

DETAILED DESCRIPTION:
Self-awareness is markedly impaired in severe mental illness including schizophrenia and schizoaffective disorder. This impairment spans awareness of symptoms as well as deficits in the estimation of abilities and capabilities, which we refer to as introspective accuracy (IA). Recent work has provided evidence of IA deficits in schizophrenia spectrum disorders, specifically in the abilities to retrospectively judge everyday functioning and neurocognitive impairment, as well as the ability to make correct real-time judgments of performance on neurocognitive tests.

Transcranial Direct Current Stimulation (tDCS) is a form of noninvasive neurostimulation which has been proposed as a therapeutic procedure in numerous psychiatric disorders. TDCS in healthy adults has been demonstrated to improve cognitive and memory performance, and in schizophrenia, tDCS has been found to improve emotion recognition ability. TDCS thus appears to be a promising therapeutic technique that may be useful for improving IA. This study will compare IA performance in individuals with schizophrenia across two conditions: active anodal tDCS and sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55
* DSM-IV-TR or DSM-5 diagnosis of schizophrenia or schizoaffective disorder and clinically stable (i.e., no hospitalizations) for at least 8 weeks and on a stable medication regimen for at least 6 weeks with no dose changes for a minimum of 2 weeks

Exclusion Criteria:

* Presence or history of pervasive developmental disorder (e.g., autism) or mental retardation (defined as IQ <70) by DSM-IV criteria
* Presence or history of medical, cardiac, or neurological disorders that may affect brain function (e.g., cardiac disease, endocrine disorders, renal disease, pulmonary disease, history of seizures or head trauma with unconsciousness for a period of 15 minutes or greater or CNS tumors)
* Presence of sensory limitation including visual (e.g., blindness, glaucoma, vision uncorrectable to 20/40) or hearing (e.g. hearing loss) impairments that interfere with assessment
* Not proficient in English
* Presence of substance abuse in the past one month
* Presence of substance dependence not in remission for the past six months
* Contraindications for tDCS (e.g., pregnancy or implanted devices such as pace maker)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pinkham, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The Unversity of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Anodal tDCS First, Then Sham Stimulation: Active anodal tDCS followed by behavioral testing; Washout (1 week); Sham stimulation followed by behavioral testing
  Intervention: Device: active anodal tDCS
- Sham tDCS First, Then Active Stimulation: Sham tDCS followed by behavioral testing; Washout (1 week); Active Stimulation followed by behavioral testing
  Intervention: Device: sham tDCS
Period: Overall Study
Arm/Group | Active Anodal tDCS First, Then Sham Stimulation | Sham tDCS First, Then Active Stimulation
Started | 21 | 20
Completed | 21 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Anodal tDCS First, Then Sham Stimulation: Active anodal tDCS followed by behavioral testing; Washout (1 week); Sham tDCS followed by behavioral testing
  Intervention: Device: active anodal tDCS
- Sham tDCS First, Then Active Stimulation: Sham tDCS followed by behavioral testing; Washout (1 week); Active tDCS followed by behavioral testing Intervention: Device: sham tDCS
  sham tDCS: sham tDCS with behavioral tasks to assess IA
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS First, Then Sham Stimulation | Sham tDCS First, Then Active Stimulation | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.43 (11.05) | 39.58 (9.84) | 39.5 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Education [Mean (Standard Deviation); unit: years] | 12.33 (2.81) | 12.34 (1.93) | 12.34 (2.41)
Estimated IQ [Mean (Standard Deviation); unit: units on a scale] | 98.95 (11.57) | 94.26 (10.01) | 96.73 (10.98)

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Introspective Accuracy for Active vs. Sham Stimulation
Description: Neurocognitive Introspective Accuracy (IA) was assessed with the Wisconsin Card Sorting Task after both Active and Sham stimulation. The area under a type 2 ROC (receiver operating characteristic) curve was used to index IA. Values range from .5-1, with higher values indicating better IA.
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Anodal tDCS: 20 minutes of Active anodal tDCS followed by behavioral testing
- Sham tDCS: 20 minutes of Sham tDCS followed by behavioral testing
Arm/Group | Active Anodal tDCS | Sham tDCS
Number analyzed (Participants) | 40 | 40
score on a scale | .534 (.068) | .526 (.085)
Statistical Analysis 1: Comparison: Active Anodal tDCS vs Sham tDCS; The null hypothesis was that of no difference in levels of IA between Active and Sham stimulation. A paired samples t-test was performed with a significance level of 0.05 (two-tailed); Test type: Superiority; p = .56, t-test, 2 sided

2. Secondary Outcome: Social Cognitive Introspective Accuracy for Active vs. Sham Stimulation
Description: Social Cognitive Introspective Accuracy assessed with the Penn Emotion Recognition Task (ER40) after both Active and Sham stimulation. The area under a type 2 ROC (receiver operating characteristic) curve was used to index IA. Values range from .5-1, with higher values indicating better IA.
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Anodal tDCS | Sham tDCS
Number analyzed (Participants) | 40 | 40
score on a scale | .575 (.095) | .562 (.098)
Statistical Analysis 1: Comparison: Active Anodal tDCS vs Sham tDCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .38, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 days after each arm.
Arm/Group | Active Anodal tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03370341/Prot_SAP_001.pdf